CLINICAL TRIAL: NCT02490917
Title: Randomised Comparative Prospective Study of the Treatment of Female Stress Urinary Incontinence Due to Intrinsic Sphincter Deficiency : ACT™ Balloon Versus Artificial Urinary Sphincter ( AMS800™)
Brief Title: ACT™ Balloons Versus Artificial Urinary Sphincter (AMS800™) for the Treatment of Female Stress Urinary Incontinence
Acronym: SU-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P130941
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Urinary Incontinence
Keywords: Female urinary incontinence; Sphincter deficiency
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT™ device (Experimental): Patients randomized to receive the Adjustable Continence Therapy device ACT™
  Interventions: Device: ACT™ device
- AMS 800 ™ device (Other): Patients randomized to receive the artificial urinary sphincter AMS 800 ™
  Interventions: Device: AMS 800 ™ device

INTERVENTIONS:
Device: ACT™ device — Implantation of the Adjustable Continence Therapy device ACT®
  Arms: ACT™ device
Device: AMS 800 ™ device — Implantation of the artificial urinary sphincter AMS 800 ™
  Arms: AMS 800 ™ device

SUMMARY:
The main objective is to compare the efficacy of AMS800 ™ and ACT ™ devices for the Treatment of Female Stress Urinary Incontinence due to Intrinsic Sphincter Deficiency on "social continence" at 6 months.

Continence is defined by the average number of pads used per day. The social continence is defined by (0-1) pad per day

DETAILED DESCRIPTION:
Prospective multicenter randomized controlled trial comparing two parallel arms: the implantation of an adjustable balloon (experimental arm) versus implantation of an artificial urinary sphincter AMS800 ™ (control arm), for the treatment of female stress urinary incontinence (SUI) due to intrinsic sphincter deficiency (ISD).

This research will focus on the assessment of improved continence, quality of life, and Cost-Effectiveness Analysis.

The tested device ACT ™ device is a prosthesis used to support the bladder neck and proximal urethra increasing the urethral coaptation and supporting to the bladder neck to prevent urine leakage at stress.

The medical device AMS 800 ™(control arm) is an implantable device made of silicone elastomer filled with saline/X-Ray fluid, used in the treatment of stress urinary incontinence related to ISD. It is designed to restore the natural process of urinary control. The device simulates normal sphincter function by closing the urethra and allowing the patient to void according to the patient's will and opening of the device (sub-cutaneous pump).

An inclusion visit will take place between 3 months and 1 month before the date of the surgery to explain the purpose of the study, the benefits and risks for patients, and describe the comparative medical devices.

Patients will be randomized before surgery (at D0).

The follow-up will be conducted up to one year, with scheduled visits at M1, M3, M6 and M12.

Secondary endpoints will be assessed during scheduled visits.

The medico-economic assessment will be made during the same follow-up period. This period will take into account improvement of urinary continence and results reported from the 3rd month as well as the morbidity and mortality related to the implementation of the medical device up to 1 year.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stress urinary incontinence due to ISD.
* Patients with maximum urethral closure pressure(PCUM) < 50 cm H2O or bladder leakage pressure < 100 cm H2O
* Patient who accepted surgery
* Patient with normal urethra-cystoscopy (no foreign body nor calculus)
* Patient with effort leaks on clinical examination
* Patient who never had SUA or ACT ™ balloon
* Affiliation to health insurance
* Written informed consent

Exclusion Criteria:

* Patient pregnant or breastfeeding
* Patient with a life expectancy of less than 2 years
* Patient with overactive bladder uncontrolled and considered an against-indication for surgery
* Patient with reduced bladder compliance
* Patient with significant post-void residual volume according to the judgment of the Investigator
* Patient with a history of pelvic radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Social continence defined by the use of 0-1 adult protective pads per day | 6 months

SECONDARY OUTCOMES:
Assessment of incontinence (number and type of protective pads used per day) | 12 months
impact on quality of life assessed by EQ-5D Health Questionnaire. | 12 months
assessment of the urinary flow using ICIQ-FLUTS questionnaire | 12 months
Assessment of Urinary Profile Symptoms using UPS questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: CHARTIER-KASTLER EMMANUEL, MD, PhD, Principal Investigator — Urology Department, Pitié-Salpêtrière University Hospital, 75013 Paris, France
Locations (1):
- Urology Department, Pitié-Salpêtrière University Hospital, Paris, France